CLINICAL TRIAL: NCT02271399
Title: Randomized Controlled Study on the Prophylaxis of Venous Thromboembolic Events in Patients Undergoing Total Knee Arthroplasty: Comparison of Aspirin and Rivaroxaban
Brief Title: Comparative Study of Prophylactic Agent for Venous Thromboembolism After Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hanyang University Seoul Hospital (Other)
Responsible Party: Principal Investigator, JIN KYU LEE, clinical assistant professor, Hanyang University Seoul Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TKRPROVTE
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Venous Thromboembolism
Keywords: venous thromboembolism; total knee arthroplasty
MeSH Terms: conditions — Venous Thromboembolism | interventions — Aspirin; Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acetylsalicylic acid (Active Comparator): aspirin 300mg tablet by mouth, every 24 hours for postoperatively 10 days
  Interventions: Drug: acetylsalicylic acid
- rivaroxaban (Experimental): xarelto 10mg tablet by mouth, every 24 hours for postoperatively 10 days
  Interventions: Drug: rivaroxaban

INTERVENTIONS:
Drug: acetylsalicylic acid — 300 mg aspirin(acetylsalicylic acid, AA, Bayer)/day was given orally for 10 days postoperatively.
  Other Names: Aspirin(Bayer)
  Arms: acetylsalicylic acid
Drug: rivaroxaban — xarelto 10mg(rivaroxaban, AA, Bayer)/day was given orally for 10 days postoperatively
  Other Names: xarelto(bayer)
  Arms: rivaroxaban

SUMMARY:
The purpose of this study is to compare the efficacy of two prophylactic agent(aspirin 300mg/day and rivaroxaban 10mg/day) for venous thromboembolism after total knee arthroplasty.

DETAILED DESCRIPTION:
1. Thromboprophylactic regimens Aspirin®(acetylsalicylic acid, AA, Bayer) 300mg/day or Xarelto® (rivaroxaban, factor Xa-inhibitor, Bayer) 10mg/day will be randomly(according to the sequence of operation) administrated in oral route to the patients undergone primary total knee replacement during postoperatively 10 days. Prophylaxis will be started at 6 hours after the end of surgery. For all patients, intermittent pneumatic compression will be initiated immediately after surgery, and a continuous passive motion machine was applied at 1 day postoperatively.
2. Evaluation and treatment plan of a VTE event

   Investigators will assess the patients for VTE(venous thromboembolism) by using a 64-channel multidetector-row computed tomography (MDCT) indirect venography system (Brilliance 64®, Philips, Eindhoven, Netherlands) at 10 days postoperatively. Six seconds after the reached 100 HU (Hounsfield units), a CT scan was performed from the costophrenic angle to the lung apex, to obtain arterial phase images of the pulmonary artery. Approximately 140 mL of contrast media (Ultravist 370®, Iopromide, Bayer) was administered through the antecubital vein at a flow rate of 4 mL/s. At 140 seconds after the injection of contrast media, indirect venography was performed from the liver dome to the ankle to obtain contrast-enhanced venous phase images. Indirect venography images were reconstructed with a slice width of 1 mm and an increment of 0.5 mm. A single radiologist evaluated the CT images in a blinded manner. Symptomatic PE was defined as PE with additional symptoms, such as dyspnea, pleuritic chest pain, cough, hemoptysis, tachypnea, rales, or tachycardia [26]. Symptomatic DVT was defined as DVT involving discomfort of the calf or thigh, a Homan's sign, swelling, localized hotness, skin discoloration, tenderness, or prominence of the superficial veins [30]. If the patient presented symptoms of those mentioned above severely, we performed MDCT before 10 days postoperatively. The VTE cases were divided into PE and DVT, and further subcategorized into proximal DVT (occurring in the popliteal vein and above) and distal DVT (occurring below the popliteal vein).

   If the patient had asymptomatic distal DVT, the patient was only observed conservatively, without any treatment. We only treated patients with PE, symptomatic DVT, or proximal DVT, and a pulmonologist or a chest surgeon was consulted for the management of these patients with anticoagulants. At 3 months postoperatively, patients who had VTE events underwent follow-up MDCT to evaluate the change in VTE.
3. Sample size assessment/Statistical analysis A power analysis was conducted prior to recruit of the patients. With prevalence of DVT postulated to be 2.94% in rivaroxaban group and 16.36% for the aspirin group after TKA, the calculation showed that 78 cases would be needed in each group to reach an alpha value of 0.05 and a confidence level of 80%.

Statistical analysis was performed with SPSS® version 18.0 for Windows (SPSS Inc, Chicago, IL, USA). For categorical variables, the Chi-square test was used to compare VTE proportions between different groups. If more than 20% of the expected frequencies were less than 5, the Fisher's exact test was performed. Moreover, one-way analysis of variance was used to compare the results of numerical continuous variables. However, for some variables without normal distribution, the Kruskal-Wallis test was used instead.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergone primary total knee arthroplasty

Exclusion Criteria:

* renal insufficiency, contrast allergy, simultaneous bilateral TKA, hemorrhagic disorder, sever liver disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
venous thromboembolism | posteropertively 10days
  Investigators evaluated the incidence of venous thromboembolism, including proximal and distal deep vein thrombosis, pulmonary embolism

SECONDARY OUTCOMES:
bleeding tendency | 2 days
  The bleeding amount was evaluated as total bleeding, which included external bleeding (drain removed routinely after 48 hours) and estimated internal bleeding (insensible loss), which was evaluated based on the method described by the Mercuriali and Inghilleri method; the preoperative estimated blood volume was calculated by Nadler's formula [20].
  Bleeding events were classified as major or minor. Major bleeding comprised intracranial, intraocular, retroperitoneal, intraspinal or pericardial bleeding . Minor bleeding included any unexpected hematoma (>25 cm2), threatened wound hematoma, nasal, gingival, rectal or vaginal bleeding, macroscopic hematuria, coughing or vomiting blood. At 10 days postoperatively, the characteristics of the bruise was assessed by using a visual analogue scale comprising 4 grades: 0 point, no bruise; 1 point, bruise limited to around the wound; 2 points, bruise extending on the calf or thigh; 3 points, bruise threatening wound healing.

CONTACTS AND LOCATIONS:
Overall Officials: Choonghyoek Choi, Study Chair — Hanyang University
Locations (1):
- Department of Orthopaedic Surgery, Hanyang University, College of Medicine, Seoul, South Korea